CLINICAL TRIAL: NCT00740168
Title: Analysis of Retinal Vessel Reaction and Monitoring of Circulation Parameters During Bevacizumab Therapy
Brief Title: Bevacizumab Treatment and Retinal Vessel Monitoring
Acronym: BevaRet
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: B-ANF1
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: bevacizumab; cancer
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TG: Bevacizumab treatment group with metastasized cancer
  Interventions: Drug: bevacizumab treatment

INTERVENTIONS:
Drug: bevacizumab treatment — single infusion 10 mg/kg
  Other Names: Avastin; ATC code: L01XC07; CAS Registry Number:216974-75-3; VEGF-inhibitor

SUMMARY:
Bevacizumab might influence the dynamic vessel function after being administered intravenously.

DETAILED DESCRIPTION:
By monitoring different vessel and circulation parameters (e.g. dynamic retinal vessel analyzer) the study will clarify the potential hemodynamic effects of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* patients who wish and need bevacizumab treatment for underlying disease

Exclusion Criteria:

* previous bevacizumab treatment
* known eye disease, eye surgery or eye trauma in history
* myopia >-2.0 dpt
* hyperopia > +2.0 dpt.
* relevant media opacity of the lens
* acute heart disease, ischemic insult, proven coronary heart disease
* cardiac arrhythmia or vessel anomalies
* seizure disorder or episode in history
* migraine
* treatment with corticosteroids within 4 weeks before study inclusion
* intake of vasoactive drugs like AT-1 or glitazone
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with first bevacizumab treatment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Diameter of retinal vessels and dynamic vessel reaction | Measurements before and after administration

SECONDARY OUTCOMES:
Baroreflex sensitivity, heart frequence variability, reaction to handgrip test | Measurements before and after administration

CONTACTS AND LOCATIONS:
Overall Officials: Tjalf Ziemssen, MD, Principal Investigator — Neurological University Clinic
Locations (1):
- Autonomic lab (ANF), Dresden, Saxony, Germany

REFERENCES:
- [Derived] Reimann M, Folprecht G, Haase R, Trautmann K, Ehninger G, Reichmann H, Ziemssen F, Ziemssen T. Anti-Vascular endothelial growth factor therapy impairs endothelial function of retinal microcirculation in colon cancer patients - an observational study. Exp Transl Stroke Med. 2013 May 13;5(1):7. doi: 10.1186/2040-7378-5-7. PMID 23668549